CLINICAL TRIAL: NCT03356769
Title: A Placebo-controlled Study of Efficacy & Safety of Aspirin as an add-on Treatment in Patients With Tuberous Sclerosis Complex (TSC) & Refractory Seizures
Brief Title: Aspirin as an add-on Treatment of Refractory Epilepsy in Tuberous Sclerosis Complex
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Shijiazhuang Yiling Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS-1425
Record Dates: First submitted 2017-11-02; First posted 2017-11-29 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2019-09

CONDITIONS: Tuberous Sclerosis Complex; Aspirin; Epilepsy; Cognitive Decline; Skin Lesions
Keywords: refractory seizure; cognitive impairment; electroencephalography improvement; seizure reduction; seizure free; aspirin
MeSH Terms: conditions — Tuberous Sclerosis; Epilepsy; Cognitive Dysfunction; Seizures | interventions — Aspirin; Anticonvulsants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, investigators, site personnel, and the sponsor's study team were masked to treatment allocation, but allocation was not concealed from personnel in charge of drug supply, and implementation of the randomisation list. The Data Safety Monitoring Board (DSMB) independent statistician and programmer were semi-blind to treatment allocation at the time of DSMB meetings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental：asprin & AEDS (Experimental): Aspirin 5mg/kg，maximum 300mg; once a day plus AEDS
  Interventions: Drug: Aspirin; Drug: AED
- control: placebo & AEDS (Placebo Comparator): placebo 5mg/kg，maximum 300mg; once a day plus AEDS
  Interventions: Drug: AED; Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — low-dose of aspirin, 5mg/Kg/d, once every day, 25mg per tablets
  Other Names: acetylsalicylic acid; enteric-coated aspirin tablets
  Arms: experimental：asprin & AEDS
Drug: AED — maintain the dosages and the drugs throughout the 3-month observation time
  Other Names: antiepileptic drugs
Drug: Placebo — placebo, 5mg/Kg/d, once every day, 25mg per tablets
  Other Names: Placebo tablets
  Arms: control: placebo & AEDS

SUMMARY:
There had been much evidence in aspirin controlling tumorous conditions conducted by basic researches, especially through mammilian target of rapamycin (mTOR) pathway. The investigator observed efficacy of aspirin in the treatment of tuberous sclerosis complex (TSC) in one child who got Kawasaki disease and in the addition four TSC patients with epilepsy. The investigator intend to evaluate whether aspirin would be an effective add-on treatment in TSC patients with refractory seizures.

DETAILED DESCRIPTION:
There is no optional treatment for patients with tuberous sclerosis complex (TSC) and refractory epilepsy.The investigator observed efficacy of aspirin in the treatment of in one child who got Kawasaki disease. Subsequent adjunctive aspirin therapy in four patients yielded a reducted frequency of seizure for 51.2-89.7%. The investigator intend to evaluate whether aspirin would be an effective add-on treatment in TSC patients with refractory seizures.

Refractory epilepsy was defined as more than 8 times of epileptic events in 4 weeks at baseline, and had been given more than two antiepileptic drugs maintaining for more than 3 months.TSC patients aged 6-30 years' old would be recruited with refractory seizures and randomly assigned to two groups, aspirin and antiepileptic drugs(AEDS) group and placebo-AEDS group after written informed consent be obtained. Patients and their guardians would be instructed to record their own seizure diary on the epileptic events and report monthly.The primary outcome would be reduction of seizure frequency (measured by average seizure frequency and response rate). The secondary outcome would include seizure-free days, seizure-free rates, changes in EEG, changes of facial angiofibromas, and exposure-response relationship analysis.The study is designed as a placebo-controlled, randomized, blinded evaluation trial.

ELIGIBILITY:
Inclusion Criteria:

1. 6-30 years old TSC patients (by Gomez criteria)
2. more than 8 seizures occurred in the 4-week baseline time,with no continued seizure-free time of more than 10 days a month
3. more than two antiepileptic drugs (AED) had been administered but fail to control the situation; maintaining with 1 or more than 1 AEDS for over 2 months and intending to continue with the drugs
4. patients who had been treated with rapamycin should have been stopped for more than 3 months
5. vagus nerve stimulation (VNS) is allowed as a previous or current therapy and would maintain until the end of the trial

Exclusion Criteria:

1. Subependymal Giant Cell Astrocytoma and requires immediate surgery；
2. a history of intracranial surgery within 6 months;
3. epilepsy caused by improper use of drugs;
4. patients treated with aspirin had severe or intolerant side effects, including gastrointestinal ulcer, bleeding, aspirin allergy, and other conditions;
5. psychogenic seizures;
6. severe renal dysfunction and infection
7. pregnant women and lactating women
8. not regular follow-up
9. other: because when children and adolescents suffering from influenza or chickenpox, using aspirin may cause a rare life-threatening Reye syndrome (characterized with persistent vomiting）, should temporary withdrawal, medication needs to consult a physician before using again.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of reduction in seizure frequency | Baseline phase (week 0); Observation phase week 1（±1 days）；Observation phase week 2（±2 days）；Observation phase week 4（±3 days）d；Observation phase week 8（±7 days）；Observation phase week 12（±14 days）
  Estimated by median percentage of seizure frequency reduction and response rate comparing each group with the baseline; response rate is defined as more than 50% of reduction in seizure frequency.
  The seizure diary of individual participants would be recorded every day during the trial time by the participants and their guardians. The correct way of recording will be guided by investigator specialized in epileptic disease with discrimination of real or false seizure events.
  •seizure information was known within the same period of time (baseline or maintenance phase)

SECONDARY OUTCOMES:
Total days of seizure free | Baseline, Week 0-4, Week 4-8, Week 8-12
  Days of seizure free in a four week observation time
A mild reduction in seizure frequency | baseline, Week 12
  At least 25% of median seizure frequency reduction comparing with those in the baseline
Changes of epileptic discharges in electroencephalogram | Baseline, Week 12
  Epileptic discharge on 2-hour video electroencephalogram in frequency detected at the same lead(s) comparing with baseline
Improvement of facial angiofibromas | Baseline, Week 4, Week 8, Week 12
  We observed improvement of facial lesions concurrent with seizure control, in the size, color and number of facial angiofibromas. The improvement will be estimated by Physician's Global Assessement Overall Score (PGA, 7-grade:more than -25%, -25% to 25%, 25-50%, 50-75%, 75%-100%, 100% improvement)
Changes of cognitive condition | Baseline, Week 12
  Raven standard reasoning test
Subjective evaluation of treatment-response condition | Baseline, Week 12
  evaluated by physician/Caregiver who is familial with the patient with Physician's Global Assessement Overall Score (PGA, 7-grade:more than -25%, -25% to 25%, 25-50%, 50-75%, 75%-100%, 100% improvement ) and a two-page age-specific questionaire

OTHER OUTCOMES:
genetic analysis | Baseline, Week 12
  genotype-phenotype correlation; evaluated by severity of symptoms and treatment effects
treatment-response annotation | Baseline phase (week 0); Observation phase week 1（±1 days）；Observation phase week 2（±2 days）；Observation phase week 4（±3 days）d；Observation phase week 8（±7 days）；Observation phase week 12（±14 days）
  Charts of seizure frequency reduction on different treatment time points would show the fluctuations of treatment effects (eg. the effective time)

CONTACTS AND LOCATIONS:
Overall Officials: Qing Liu, MD PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Neurology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Franz DN, Leonard J, Tudor C, Chuck G, Care M, Sethuraman G, Dinopoulos A, Thomas G, Crone KR. Rapamycin causes regression of astrocytomas in tuberous sclerosis complex. Ann Neurol. 2006 Mar;59(3):490-8. doi: 10.1002/ana.20784. PMID 16453317
- [Background] Krueger DA, Care MM, Holland K, Agricola K, Tudor C, Mangeshkar P, Wilson KA, Byars A, Sahmoud T, Franz DN. Everolimus for subependymal giant-cell astrocytomas in tuberous sclerosis. N Engl J Med. 2010 Nov 4;363(19):1801-11. doi: 10.1056/NEJMoa1001671. PMID 21047224
- [Background] Din FV, Valanciute A, Houde VP, Zibrova D, Green KA, Sakamoto K, Alessi DR, Dunlop MG. Aspirin inhibits mTOR signaling, activates AMP-activated protein kinase, and induces autophagy in colorectal cancer cells. Gastroenterology. 2012 Jun;142(7):1504-15.e3. doi: 10.1053/j.gastro.2012.02.050. Epub 2012 Mar 6. PMID 22406476
- [Background] Chen CT, Du Y, Yamaguchi H, Hsu JM, Kuo HP, Hortobagyi GN, Hung MC. Targeting the IKKbeta/mTOR/VEGF signaling pathway as a potential therapeutic strategy for obesity-related breast cancer. Mol Cancer Ther. 2012 Oct;11(10):2212-21. doi: 10.1158/1535-7163.MCT-12-0180. Epub 2012 Jul 23. PMID 22826466
- [Background] Northrup H, Krueger DA; International Tuberous Sclerosis Complex Consensus Group. Tuberous sclerosis complex diagnostic criteria update: recommendations of the 2012 Iinternational Tuberous Sclerosis Complex Consensus Conference. Pediatr Neurol. 2013 Oct;49(4):243-54. doi: 10.1016/j.pediatrneurol.2013.08.001. PMID 24053982
- [Background] Overwater IE, Rietman AB, Bindels-de Heus K, Looman CW, Rizopoulos D, Sibindi TM, Cherian PJ, Jansen FE, Moll HA, Elgersma Y, de Wit MC. Sirolimus for epilepsy in children with tuberous sclerosis complex: A randomized controlled trial. Neurology. 2016 Sep 6;87(10):1011-8. doi: 10.1212/WNL.0000000000003077. Epub 2016 Aug 10. PMID 27511181
- See also: Rapamycin in TSC — https://www.ncbi.nlm.nih.gov/pubmed/?term=Franz%2C+D.N.%2C+et+al.%2C+Rapamycin+causes+regression+of+astrocytomas+in+tuberous+sclerosis+complex.+Ann+Neurol%2C+2006.+59(3)%3A+p.+490-8.
- See also: Rapamycin in TSC — https://www.ncbi.nlm.nih.gov/pubmed/?term=Krueger%2C+D.A.%2C+et+al.%2C+Everolimus+for+subependymal+giant-cell+astrocytomas+in+tuberous+sclerosis.+N+Engl+J+Med%2C+2010.+363(19)%3A+p.+1801-1
- See also: basic study on aspirin-mTOR — https://www.ncbi.nlm.nih.gov/pubmed/?term=Din%2C+F.V.%2C+et+al.%2C+Aspirin+inhibits+mTOR+signaling%2C+activates+AMP-activated+protein+kinase%2C+and+induces+autophagy+in
- See also: basic study on aspirin-mTOR — https://www.ncbi.nlm.nih.gov/pubmed/?term=Targeting+the+IKKbeta%2FmTOR%2FVEGF+signaling+pathway+as+a+potential+therapeutic+strategy+for+obesity-related+breast+cancer.+Mol+Cancer+Ther%2C+2012.+11(10)%3A+p.+2212-21
- See also: TSC — https://www.ncbi.nlm.nih.gov/pubmed/?term=International+Tuberous+Sclerosis+Complex+Consensus%2C+Tuberous+sclerosis+complex+diagnostic+criteria+update%3A+recommendations+of+the+2012+Iinternational+Tuberous+Sclerosis+Complex+Consensus+Conference.
- See also: Rapamycin in TSC — https://www.ncbi.nlm.nih.gov/pubmed/27511181